CLINICAL TRIAL: NCT03594240
Title: The Role of Vitamin B Complex as an Adjuvant Therapy for Diabetic Nephropathy in Pediatric Patients With Type 1 Diabetes
Brief Title: Vitamin B Complex and Diabetic Nephropathy in Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nancy Samir Elbarbary, Professor of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ain Shams Pediatrics 2082016
Record Dates: First submitted 2018-06-30; First posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Plasma Homocysteine; HbA1c Level
MeSH Terms: interventions — Vitamin B Complex

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned into two groups; intervention group who received vitamin B complex once daily orally and control group who did not receive B complex
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): Intervention group included pediatric patients with diabetic nephropathy receiving oral vitamin B complex tablets( Neurorubine TM -Forte Lactab TM ) once daily.
  Interventions: Drug: Vitamin B complex tablets (Neurorubine TM -Forte Lactab TM)
- Control group (Placebo Comparator): Placebo group or control patients received placebo that were similar in appearance to vitamin B complex tablets and the administered dose was as the same schedule as vitamin B complex .
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Drug: Vitamin B complex tablets (Neurorubine TM -Forte Lactab TM) — Vitamin B complex tablets (Neurorubine TM -Forte Lactab TM) once daily
  Arms: intervention group
Dietary Supplement: Placebo — Patients in placebo group received placebo that were similar in appearance to Vitamin B complex tablets and the administered dose was as the same schedule as Vitamin B complex.
  Arms: Control group

SUMMARY:
Homocysteine levels have been found elevated in T1DM patients with Diabetic nephropathy (DN) due to several causes, including dietary deficiencies. Hyperhomocysteinemia induces renal injury and is associated with increasing urinary albumin excretion(UAE). Therefore, the investigators performed a randomized-controlled trial of oral supplementation with vitamin B complex as an adjuvant therapy for nephropathy in pediatric patients with T1DM and assessed its relation to homocysteine levels, glycemic control, microalbuminuria and cystatin C as a marker of nephropathy.

DETAILED DESCRIPTION:
This trial included 80 vitamin B12-deficient T1DM patients with nephropathy, despite oral angiotensin-converting enzyme inhibitors . Enrolled patients aged 12-18 years with at least 5 years disease duration and HbA1c ≤8.5%. Patients were randomly assigned into two groups; intervention group who received vitamin B complex once daily orally . The other group did not receive any supplementation and served as a control group. Both groups were followed-up for 12 weeks with assessment of plasma homocysteine, HbA1c, cystatin C and UAE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes.
* Patients aged 12-18 years with at least 5 years disease duration.
* Active diabetic nephropathy in the form of microalbuminuria (urinary albumin excretion [UAE] 30-299 mg/g creatinine in two of three samples over a 3- to 6- months period despite angiotensin converting enzyme inhibitors)
* Hemoglobin A1c (HbA1c) ≤8.5%
* Patients on regular visit to clinic.
* Patients on regular insulin therapy.

Exclusion Criteria:

Patients were excluded if they have any of the following:

* Patients with history of liver disease or any disorder likely to impair liver functions or elevated liver enzymes.
* Patients with any evidence of renal impairment due to cause other than diabetes.
* Patients with hypertension.
* Hepatitis virus infection (B or C) or any evidence of infection.
* Taking any vitamins or food supplements one month before study.
* Participation in a previous investigational drug study within 3 months preceding screening.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Change in plasma homocysteine | 12 weeks
  Change in plasma homocysteine level after 12 weeks of oral vitamin B complex intake

SECONDARY OUTCOMES:
Change in HbA1c level | 12 weeks
  Change in HbA1c level after 12 weeks of oral vitamin B complex intake

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy Elbarbary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Mainly clinical characteristics

REFERENCES:
- [Derived] Elbarbary NS, Ismail EAR, Zaki MA, Darwish YW, Ibrahim MZ, El-Hamamsy M. Vitamin B complex supplementation as a homocysteine-lowering therapy for early stage diabetic nephropathy in pediatric patients with type 1 diabetes: A randomized controlled trial. Clin Nutr. 2020 Jan;39(1):49-56. doi: 10.1016/j.clnu.2019.01.006. Epub 2019 Jan 17. PMID 30704890